## **Statistical Analysis Plan**

Official Title: Comparison of Total Intravenous Anesthesia Methods in Patients Undergoing

Neuromonitoring

**NCT Number:** Pending (Not yet assigned)

**Document Date:** May 10, 2023

## **Statistical Analysis:**

Statistical analyses were performed using SPSS (IBM SPSS Statistics 27). Patients were grouped based on the TIVA protocol applied:

• **Group S:** Propofol and remifentanil (n=24)

• **Group K:** Propofol, remifentanil, and ketamine (n=24)

• **Group L:** Propofol, remifentanil, and lidocaine (n=24)

For normally distributed data, parametric tests were used:

• Independent Samples t-test for comparing two groups.

• ANOVA for comparing three or more groups.

For non-normally distributed data, non-parametric tests were applied:

- Mann-Whitney U for two-group comparisons.
- Kruskal-Wallis H for comparisons of three or more groups.

Post-hoc pairwise comparisons with Bonferroni correction were performed for variables with significant differences.